CLINICAL TRIAL: NCT03155607
Title: Novel Virtual Reality for Burn Wound Care Pain in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 206406
Record Dates: First submitted 2017-05-12; First posted 2017-05-16 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention)
- Virtual Reality Distraction (Experimental)
  Interventions: Behavioral: Virtual Reality Distraction

INTERVENTIONS:
Behavioral: Virtual Reality Distraction — Patient will utilize a virtual reality device during wound care.
  Arms: Virtual Reality Distraction

SUMMARY:
Burn wounds cause intense, complex pain, and subsequent burn wound care causes further intense, episodic pain that is often unrelieved by opioid and non-opioid medications, resulting in under-treatment of pain. Further, opioid analgesics can have untoward side effects including respiratory depression, nausea, constipation, pruritus, drowsiness, lethargy, dependence, and induced hyperalgesia. As one of the most severe types of pain, burn wound care pain adds to the trauma pediatric patients already experience from the burn itself impacting quality of life with subsequent behavioral and maladaptive responses, such as agitation, anger, anxiety, hyperactivity, uncooperativeness, aggression, and dissociation. Lack of control over the procedure, pain memory, anxiety in anticipation of the repeated painful nature of the procedure, and transmission of clinician distress associated with inflicting procedural pain on the child contribute to the pain perceived.

Virtual reality (VR) shows great promise as an engaging, interactive, effective non-pharmacologic intervention for various painful healthcare procedures, including burn wound care, therapies, and chronic pain conditions, despite equivocal findings, perhaps due to methodological issues. Designs of many studies of VR during burn wound care have been case studies or carefully controlled within-subject designs; sample sizes have been small. Recommendations for ongoing research include conducting more rigorous studies including randomized controlled trials (RCTs), repeat design studies, testing VR throughout the healthcare procedure, comparing VR to other distraction interventions; and using larger sample sizes.

Primary Aim 1: Compare the effectiveness of age-appropriate, consumer available, high technology, interactive VR with standard care (SC) on adolescents' acute procedural pain intensity perception during burn wound care treatment in the ambulatory outpatient clinic setting.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing burn wound care
* First visit to the outpatient Arkansas Children's Hospital (ACH) Burn Clinic or first wound care procedure in the Burn Clinic without sedation
* Ages 10 through 21 years (based on a developmental framework of early adolescence: 10-13 years, middle-adolescence: 14-17 years, and late adolescence: 18-21 years)
* English speaking (Note: Not all data collection tools are available in languages other than English)

Exclusion Criteria:

* Any wounds that may interfere with study procedures (Previously, we did not have to exclude facial, head, neck or hand burns but were able to adapt the VR equipment.)
* History of motion sickness, seizure disorder, dizziness, or migraine headaches precipitated by visual auras
* Incarcerated minors
* Minors in foster care
* Presence of a cognitive developmental disability determined on prescreening by presence of a Section 504 accommodation plan or Title VIII individualized educational plan (IEP) in school. If IEP or 504 plan is unrelated to a cognitive delay, then the adolescent will be included in the study.

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2021-12-02 (Actual)

PRIMARY OUTCOMES:
Pain perception during burn wound care of first clinic visit | From study consent, data collection, and randomization at beginning of clinic visit until final data collection at discharge from clinic; approximately 2 hours.
  Pain perception as described by utilizing the Adolescent Pediatric Pain Tool. Pain is based on a 0 (No pain) to 10 (maximum pain) sonometer scale as told by patient

CONTACTS AND LOCATIONS:
Overall Officials: Debra Jeffs, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No